CLINICAL TRIAL: NCT00880204
Title: Evaluation of Essential Surgical Skills-Emergency Maternal and Child Health (ESS-EMCH) Training by Assessing the Doctors' Practices in Pakistan
Brief Title: Evaluation of Essential Surgical Skills-Emergency Maternal and Child Health Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Child Advocacy International (Other)
Collaborators: John Snow, Inc. (Industry); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Yasir Bin Nisar, Researcher, Child Advocacy International
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CRT2008
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Sepsis; Asthma; Heart Failure; Seizure; Coma
Keywords: Cluster Randomized Trial; ESS-EMCH; Neonatal; Maternal; Life threatening emergency event
MeSH Terms: conditions — Sepsis; Asthma; Heart Failure; Seizures; Coma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trained doctors (Experimental): ESS-EMCH Training will be provided to doctors working in general emergency, pediatrics and obstetrics department in district hospitals.
  Interventions: Behavioral: ESS-EMCH training
- No Training (No Intervention): No training will be given to doctors (act as controls)

INTERVENTIONS:
Behavioral: ESS-EMCH training — The trainings of the ESS-EMCH programme are based on two well-tried and tested structured training methodologies of "Advanced Pediatric Life Support (APLS)" and "Management of Obstetric Emergencies and Trauma (MOET)".
  Arms: Trained doctors

SUMMARY:
The aim of the proposed study is to determine if specific training in management of general, obstetric, neonatal and pediatric emergencies results in a change in practice of doctors working in emergency departments of public sector hospitals in three districts of Pakistan. The overall goal of the proposed study is to test the ability of a standard course (5-days training) to promote the provision of effective and evidence based practices in public sector hospital settings.

DETAILED DESCRIPTION:
Pakistan is the 6th most populous country of the world 1 and has the largest population in the Eastern Mediterranean Region, accounting for about 30 percent of the regional population. The level of socio-economic development is still low - GDP per capita is US$ 7302; HDI is 142nd in the world 1; and, one fourth of the entire population lives below the poverty line 2. The health profile of Pakistan is characterized by high population growth rate, high infant and child mortality rate, high maternal mortality ratio, and high burden of communicable diseases.

In conjunction with neonatal, infant and child mortality, maternal mortality ratio is also extremely high as 350 per 100,000 population in Pakistan 3. In addition, only 23 percent of the deliveries are being conducted by skilled birth attendants and major causes of mortality include hemorrhage, hypertensive diseases, sepsis and other obstetrical complications 4. Although the health facilities are available ubiquitously, but these facilities lack proper equipments and trained health workers. Health worker also lacks necessary skills and training to manage the children, newborns and mothers in emergency situations. Management in the first few hours - the Golden hours 5 of the presentation of obstetric, neonatal and pediatric emergencies, including major trauma (if not given immediate attention are likely to result in death or severe brain damage in 6 hours) is a major determinant of the eventual outcome. If the vast majority of these potentially avoidable deaths and long-term or permanent morbidity are to be avoided, a continuity of care with particular emphasis on golden hours management and safe transfer has to be established starting from the communities to health facilities 6.

There is evidence that if structured life support trainings are introduced in a systematic method it helps in reducing mortality and morbidity during the emergency phase in a very cost effective manner 4. Local public sector hospitals need to be configured to serve a community and not just to provide episodic care for the few patients who transiently pass through their doors during an acute episode. It is mandatory to upgrade the knowledge of first line health worker in managing emergency situations. It is also necessary to elevate their capacity to recognize the common emergencies and manage accordingly. By instituting accredited structured training for these skills we can dramatically decrease mortality and morbidity rates in Pakistan 6. The training activities of Essential Surgical Skills with emphasis on Emergency Maternal and Child Health (ESS-EMCH) are based on two tried and tested structured training methodologies of Advanced Pediatric Life Support (APLS) and Management of Obstetric Emergencies and Trauma (MOET). The ESS-EMCH training programme is being conducted by Child Health Advocacy International (CAI) in Pakistan and Gambia 6. The Advanced Life Support Group-UK (ALSG-UK) and World Health Organization (WHO) provide technical support for the training and the programme has been endorsed as a first ALSG-UK certified training course targeted specifically for developing countries 7. These courses have been used for some years in various developed countries as essential requirements for all health workers involved in emergency care in these specialties. In Pakistan these training activities have been modified according to local needs and conditions 6.

The aim of the proposed study is to determine, if and what degree, specific training in management of general, obstetric, neonatal and pediatric emergencies results in a change in practice of doctors working in emergency departments of public sector hospitals in three districts of Pakistan. The overall goal of the proposed study is to test the ability of a standard course (5-days training) to promote the provision of effective and evidence based practices in public sector hospital settings.

Justification:

Improving mortality and morbidity during the emergency phase presents a major challenge in many developing countries including Pakistan. It is important that health workers working at public health facilities at district level have necessary skills and equipment to provide effective management during an emergency phase. Research has shown that structured life support trainings can help in reducing mortality and morbidity during the emergency phase in a very cost effective manner 4. However, the evaluation of course participants poses a major problem, because it is rarely possible to develop a perfect testing method, and awareness of the inherent limitations of evaluation methods used in life support courses is important 8. Jabbour and colleagues reviewed the effectiveness of life support courses and found that the majority of studies on evaluation of the ability of life support courses have focused on less direct outcomes like health workers' knowledge and silks 9. Such surrogate outcomes may not necessarily reflect practice changes, which is a more useful and direct way of measuring the effectiveness of life support training courses 9.

We are not aware of any previous randomized controlled trials determining the effect of ESS-EMCH training on health workers practices in a true clinical setting. Therefore, our intention is to test the ability of ESS-EMCH training on practices by randomly assigning pediatric ward, labor room and emergency department staff at district level to either providing ESS-EMCH training or no training, considering the health worker as a unit of cluster. Although, our primary outcome will only able to capture the initial steps in effective practice, but we believe it will indicate an important behavior change effect.

ELIGIBILITY:
Inclusion Criteria:

* doctors working in emergency department, pediatrics and obstetric department in district hospitals

Exclusion Criteria:

* doctors at leave for more than 1 week
* working in other departments of district hospitals

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2009-09-30 (Actual); Study Completion 2009-11-30 (Actual)

PRIMARY OUTCOMES:
To examine the ability of ESS-EMCH to change doctors' practices for managing obstetric, neonatal, and pediatric emergency care, including major trauma, in public sector hospital settings | 1-2 months
  Practices

CONTACTS AND LOCATIONS:
Overall Officials: Yasir B Nisar, MPH, Principal Investigator — CAI
Locations (2):
- Pakistan (2):
  - CAI, Islamabad, Capital
  - District Headquarters Hospital, Vehari, Punjab Province